CLINICAL TRIAL: NCT06900010
Title: An Open-label, Dose Escalation Phase Ⅰ/Ⅱ Study to Evaluate the Efficacy and Safety of CM336 (BCMA/CD3 Bispecific Antibody) in Adults with Moderate to Severe Autoimmune Bullous Disease
Brief Title: A Study to Evaluate CM336 in Adults with Autoimmune Bullous Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM336-IIS-PP01
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Bullous Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention(CM336) (Experimental)
  Interventions: Biological: CM336 Injection

INTERVENTIONS:
Biological: CM336 Injection — subcutaneous CM336 administration

SUMMARY:
to Evaluate the Efficacy and Safety of CM336 (BCMA/CD3 Bispecific Antibody) in Adults with Moderate to Severe Autoimmune Bullous Disease

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed diagnosis of autoimmune bullous disease；
* 2. Age ≥18 years, regardless of gender；
* 3. Voluntarily signed informed consent form, with understanding of the study's nature, purpose, procedures, and willingness to comply with trial requirements.

Exclusion Criteria:

* 1. History of clinically significant diseases that, in the investigator's judgment, may pose safety risks to the subject during participation；
* 2. Prior treatment with anti-B-cell maturation antigen (BCMA) therapy；
* 3. History of allergic reactions to humanized monoclonal antibodies or known allergy to any component of CM336；
* 4. Any other condition deemed by the investigator to render the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy after CM336 treatment | Up to 52 weeks
  Proportion of subjects in remission

CONTACTS AND LOCATIONS:
Overall Officials: Furen Zhang, Principal Investigator — Dermatology Hospital affiliated to Shandong First Medical University
Locations (1):
- Dermatology Hospital Affiliated to Shandong First Medical University, Jinan, China